CLINICAL TRIAL: NCT00807248
Title: Randomised, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study of Escitalopram in Combination With Two Fixed Doses of Gaboxadol Compared to Escitalopram in Major Depressive Disorder
Brief Title: Short-term Study of Combination Treatment of Escitalopram and Gaboxadol in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12213A; 2008-000506-36 (Registry Identifier: EudraCT)
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; gaboxadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Escitalopram placebo and gaboxadol placebo (Placebo Comparator)
  Interventions: Drug: Escitalopram placebo; Drug: Gaboxadol placebo
- Escitalopram 20 mg and gaboxadol placebo (Active Comparator)
  Interventions: Drug: Gaboxadol placebo; Drug: Escitalopram 20 mg
- Escitalopram 20 mg and gaboxadol 5 mg (Experimental)
  Interventions: Drug: Escitalopram 20 mg; Drug: Gaboxadol 5 mg
- Escitalopram 20 mg and gaboxadol 10 mg (Experimental)
  Interventions: Drug: Escitalopram 20 mg; Drug: Gaboxadol 10 mg

INTERVENTIONS:
Drug: Escitalopram placebo — Once daily before bedtime for 8 weeks
  Arms: Escitalopram placebo and gaboxadol placebo
Drug: Gaboxadol placebo — Once daily before bedtime for 8 weeks
  Arms: Escitalopram 20 mg and gaboxadol placebo; Escitalopram placebo and gaboxadol placebo
Drug: Escitalopram 20 mg — Once daily before bedtime for 8 weeks
  Other Names: Escitalopram = Cipralex/Lexapro/Seroplex/Sipralexa
  Arms: Escitalopram 20 mg and gaboxadol 10 mg; Escitalopram 20 mg and gaboxadol 5 mg; Escitalopram 20 mg and gaboxadol placebo
Drug: Gaboxadol 5 mg — Once daily before bedtime for 8 weeks
  Arms: Escitalopram 20 mg and gaboxadol 5 mg
Drug: Gaboxadol 10 mg — Once daily before bedtime for 8 weeks
  Arms: Escitalopram 20 mg and gaboxadol 10 mg

SUMMARY:
To compare the efficacy of escitalopram fixed dose 20 mg/day in combination with fixed doses of gaboxadol (5 and 10 mg/day) versus escitalopram fixed dose 20 mg/day after 8 weeks of treatment in patients with Major Depressive Disorder

DETAILED DESCRIPTION:
Subjects participating in this study will be respectively randomised (1:2:2:2) to receive either:

* placebo or
* escitalopram 20 mg/day or
* escitalopram 20 mg/day in combination with gaboxadol 5 mg/day or
* escitalopram 20 mg/day in combination with gaboxadol 10 mg/day

ELIGIBILITY:
Inclusion Criteria:

Clinical Diagnosis of MDD according to DSM-IV-TR criteria:

* With reported duration of the current major depressive episode of at least 3 months
* With MADRS total score of at least 30

Exclusion Criteria:

The patient has 1 or more of the following:

* Any current psychiatric disorder other than MDD as defined in the DSM-IV-TR
* Current or past history of: manic or hypomanic episode, schizophrenia, or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR
* Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR
* Presence or history of a clinically significant neurological disorder (including epilepsy)
* Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc)
* Any Axis II disorder that might compromise the study
* Previous use of hallucinogenic drug

The patient has a significant risk of suicide according to the investigator's opinion, or has a score >=5 on item 10 (suicidal thoughts) of the MADRS, or has made a suicide attempt in the previous 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (22):
- AT001, Vienna, Austria
- Russia (21):
  - RU019, Barnaul
  - RU029, Izhevsk
  - RU020, Kemerovo
  - RU012, Krasnodar
  - RU010, Krasnodar
  - RU022, Kursk
  - RU015, Moscow
  - RU026, Moscow
  - RU001, Moscow
  - RU002, Moscow
  - RU028, Moscow
  - RU003, Moscow
  - RU007, Moscow
  - RU027, Saransk
  - RU024, Saratov
  - RU013, Saratov
  - RU021, Tomsk
  - RU016, Tver'
  - RU014, Volgograd
  - RU011, Yaroslavl
  - RU018, Yekaterinburg

REFERENCES:
- [Result] Kasper S, Ebert B, Larsen K, Tonnoir B. Combining escitalopram with gaboxadol provides no additional benefit in the treatment of patients with severe major depressive disorder. Int J Neuropsychopharmacol. 2012 Jul;15(6):715-25. doi: 10.1017/S146114571100112X. Epub 2011 Oct 19. PMID 22008735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from specialist inpatient and outpatient clinics.
Period: Overall Study
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Started | 71 | 140 | 139 | 140
Completed | 50 | 128 | 121 | 126
Not Completed | 21 | 12 | 18 | 14
Not completed — Adverse Event | 1 | 2 | 2 | 6
Not completed — Lack of Efficacy | 14 | 4 | 8 | 3
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Withdrawal of Consent | 5 | 5 | 5 | 5
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Other Reason | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily) | Total
Number analyzed (Participants) | 71 | 140 | 139 | 140 | 490
Age Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.6) | 41.6 (12.6) | 42.6 (11.8) | 41.5 (10.5) | 42.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 96 | 96 | 93 | 338
  Male | 18 | 44 | 43 | 47 | 152
Montgomery and Åsberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: Scores on a scale] — The MADRS is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at 2-point intervals. The total score of the 10 items ranges from 0 to 60.
  Scores on a scale | 34.7 (4.2) | 35.4 (4.3) | 35.3 (3.4) | 34.7 (3.8) | 35.1 (3.9)
Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: Scores on a scale] — The HADS is a patient-rated scale designed to screen for anxiety and depressive states in medical patients. It consists of two sub-scales: the D-scale measures depression and the A-scale measures anxiety. Each sub-scale contains 7 items, and each item is rated from 0 (absent) to 3 (maximum severity). The score of each sub-scale ranges from 0 to 21, and are analysed separately. The total HADS score ranges from 0 to 42.
  Scores on a scale | 27.5 (5.9) | 28.2 (5.3) | 28.1 (5.5) | 27.4 (5.5) | 27.8 (5.5)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: Scores on a scale] — The ISI is both a brief screening measure of insomnia and an outcomes measure for use in treatment research. It is a brief self-report instrument measuring the patient's perception of his or her insomnia, and it comprises 7 items. Each item is rated on a 0-4 scale and the total score ranges from 0 to 28. 0 = no symptoms and 28 = severe symptoms.
  Scores on a scale | 18.4 (5.0) | 18.6 (4.7) | 18.2 (4.4) | 18.1 (4.8) | 18.3 (4.7)
Sheehan Disability Scale (SDS): Family Subscale [Mean (Standard Deviation); unit: Scores on a scale] — The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment.
  Scores on a scale | 7.0 (1.4) | 7.1 (1.6) | 7.2 (1.3) | 6.9 (1.4) | 7.1 (1.4)
SDS: Work Subscale [Mean (Standard Deviation); unit: Scores on a scale] — The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment.
  Scores on a scale | 7.3 (1.2) | 7.4 (1.3) | 7.3 (1.5) | 7.0 (1.4) | 7.2 (1.4)
SDS: Social Subscale [Mean (Standard Deviation); unit: Scores on a scale] — The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment.
  Scores on a scale | 7.0 (1.4) | 7.1 (1.4) | 7.1 (1.5) | 6.9 (1.6) | 7.0 (1.5)
Clinical Global Impression - Severity of Illness (CGI-S) [Mean (Standard Deviation); unit: Scores on a scale] — The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
  Scores on a scale | 4.4 (0.9) | 4.5 (0.9) | 4.3 (0.9) | 4.4 (0.9) | 4.4 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery and Åsberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at 2-point intervals. The total score of the 10 items ranges from 0 to 60.
Time Frame: Baseline to 8 weeks
Population: Mean change from baseline to Week 8: Full-analysis Set (FAS), Last Observation Carried Forward (LOCF), Analysis of Covariance (ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -13.4 (1.1) | -19.0 (0.9) | -18.5 (0.9) | -19.4 (0.9)
Statistical Analysis 1: Comparison: Escitalopram 20 mg and Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p = 0.6405, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-2.34 to 1.44], Standard Error of Mean 0.96
Statistical Analysis 2: Comparison: Escitalopram 20 mg and Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p = 0.6227, ANCOVA; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-1.41 to 2.35], Standard Error of Mean 0.96

2. Secondary Outcome: MADRS
Description: as for outcome 1
Time Frame: From baseline to Week 8
Population: Mean change from baseline to Week 8 (FAS, LOCF, ANCOVA)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -13.4 (1.1) | -19.0 (0.9) | -18.5 (0.9) | -19.4 (0.9)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -5.55, 95% CI 2-sided [-7.98 to -3.11], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -5.09, 95% CI 2-sided [-7.53 to -2.66], Standard Error of Mean 1.24
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -6.00, 95% CI 2-sided [-8.43 to -3.56], Standard Error of Mean 1.24

3. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a patient-rated scale designed to screen for anxiety and depressive states in medical patients. It consists of two sub-scales: the D-scale measures depression and the A-scale measures anxiety. Each sub-scale contains 7 items, and each item is rated from 0 (absent) to 3 (maximum severity). The score of each sub-scale ranges from 0 to 21, and are analysed separately. The total HADS score ranges from 0 to 42.
Time Frame: Mean change from baseline to Week 8
Population: Mean change from baseline to Week 8 (FAS, LOCF, ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -9.7 (1.0) | -14.7 (0.8) | -14.1 (0.8) | -15.0 (0.7)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.98, 95% CI 2-sided [-7.13 to -2.84], Standard Error of Mean 1.09
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.46, 95% CI 2-sided [-6.60 to -2.32], Standard Error of Mean 1.09
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -5.27, 95% CI 2-sided [-7.41 to -3.13], Standard Error of Mean 1.09

4. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The ISI is both a brief screening measure of insomnia and an outcomes measure for use in treatment research. It is a brief self-report instrument measuring the patient's perception of his or her insomnia, and it comprises 7 items. Each item is rated on a 0-4 scale and the total score ranges from 0 to 28. 0 = no symptoms and 28 = severe symptoms.
Time Frame: Mean change from baseline to Week 8
Population: Mean change from baseline to Week 8 (FAS, LOCF, ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -6.9 (0.7) | -10.0 (0.5) | -9.6 (0.5) | -10.6 (0.5)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.09, 95% CI 2-sided [-4.59 to -1.58], Standard Error of Mean 0.77
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -2.64, 95% CI 2-sided [-4.15 to -1.14], Standard Error of Mean 0.77
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.61, 95% CI 2-sided [-5.13 to -2.10], Standard Error of Mean 0.77

5. Secondary Outcome: Sheehan Disability Scale (SDS): Family Subscale
Description: The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment.
Time Frame: Mean change from baseline to Week 8
Population: Mean change from baseline to Week 8 (FAS, LOCF, ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -2.8 (0.02) | -4.0 (0.02) | -3.9 (0.02) | -4.1 (0.02)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-1.85 to -0.64], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-1.72 to -0.50], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-1.87 to -0.65], Standard Error of Mean 0.31

6. Secondary Outcome: SDS: Work Subscale
Description: as for outcome 5
Time Frame: Mean change from baseline to Week 8
Population: Mean change from baseline to Week 8 (FAS, LOCF, ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -2.7 (0.03) | -3.8 (0.02) | -3.8 (0.02) | -4.0 (0.02)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-1.72 to -0.46], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p = 0.0013, ANCOVA; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.69 to -0.41], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-1.92 to -0.66], Standard Error of Mean 0.32

7. Secondary Outcome: SDS: Social Subscale
Description: as for outcome 5
Time Frame: Mean change from baseline to Week 8
Population: Mean change from baseline to Week 8 (FAS, LOCF, ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -2.7 (0.03) | -3.9 (0.02) | -3.8 (0.02) | -4.1 (0.02)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.82 to -0.58], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-1.72 to -0.48], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-2.00 to -0.76], Standard Error of Mean 0.32

8. Secondary Outcome: Clinical Global Impression - Severity of Illness (CGI-S)
Description: The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Mean change from baseline to Week 8
Population: Mean change from baseline to Week 8 (FAS, LOCF, ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | -1.04 (0.13) | -1.65 (0.10) | -1.58 (0.10) | -1.76 (0.10)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.89 to -0.34], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.82 to -0.26], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-0.99 to -0.44], Standard Error of Mean 0.14

9. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I)
Description: The CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: at Week 8
Population: At Week 8 (FAS, LOCF, ANCOVA)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Number analyzed (Participants) | 71 | 139 | 139 | 140
Scores on a scale | 2.97 (0.12) | 2.21 (0.09) | 2.35 (0.09) | 2.26 (0.09)
Statistical Analysis 1: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Placebo (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-1.02 to -0.50], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.88 to -0.36], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo (Orally, Once Daily) vs Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-0.97 to -0.45], Standard Error of Mean 0.13

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Placebo (Orally, Once Daily) | Escitalopram 20 mg and Placebo (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily)
Serious Adverse Events (participants affected / at risk) | 1/71 | 0/140 | 0/139 | 0/140
Other Adverse Events (participants affected / at risk) | 12/71 | 22/140 | 31/139 | 19/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Orally, Once Daily) (N=71) | Escitalopram 20 mg and Placebo (Orally, Once Daily) (N=140) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) (N=139) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily) (N=140)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Orally, Once Daily) (N=71) | Escitalopram 20 mg and Placebo (Orally, Once Daily) (N=140) | Escitalopram 20 mg and Gaboxadol 5 mg (Orally, Once Daily) (N=139) | Escitalopram 20 mg and Gaboxadol 10 mg (Orally, Once Daily) (N=140)
Headache (Nervous system disorders) | 4 | 7 | 5 | 3
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 3 | 2 | 3
Insomnia (Psychiatric disorders) | 3 | 3 | 4 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 4 | 8 | 3
Blood pressure increased (Investigations) | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 6 | 2
Dermatitis allergic (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 2
Rhinitis allergic (Infections and infestations) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub-publications.